CLINICAL TRIAL: NCT00498576
Title: Melatonin and Adiponectin in Hypertensive Kidney Transplant
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: leibowitz avshalom, Sheba Medical Center
Other Study IDs: SHEBA-07-4730-AL-CTIL
Record Dates: First submitted 2007-07-08; First posted 2007-07-10 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Hypertension; Kidney Transplant
Keywords: hypertension; kidney transplant; melatonin; adiponectin
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: kidney transplant with hypertension
- 2: hypertensive patients with native kidneys
- 3: healthy controls

SUMMARY:
Recently we have shown that melatonin secretion is impaired in rats with metabolic syndrome. We have also demonstrated that exogenic melatonin supplementation can improve blood pressure profile in nondipper patients.

The aim of this study is to find whether there is a difference between melatonin secretion in hypertensive kidney recipients versus "normal" hypertensive patients. Secondly, to ask if there is any correlation between melatonin secretion and adiponectin levels.

ELIGIBILITY:
Inclusion Criteria:

* hypertension
* kidney transplantation ( group 1)
* good renal function

Exclusion Criteria:

* diabetes mellitus
* cancer
* renal failure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: group1- patients from the kidney transplant unit, sheba medical center group2- patients from hypertension unit,sheba medical center
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2007-09

CONTACTS AND LOCATIONS:
Overall Officials: Avshalom Leibowitz, MD, Principal Investigator
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel